CLINICAL TRIAL: NCT03800147
Title: Effects of Nutritional Fat on the Growth of Intestinal E. Coli
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FAT Study
Record Dates: First submitted 2018-12-13; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Escherichia Coli Infections
MeSH Terms: conditions — Escherichia coli Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: randomized controlled crossover clinical study
Who Masked: Investigator
Masking Description: Participants will not be blinded regarding the composition of their nutrition. Investigators performing stool and blood analyses will be blinded to the group assignment of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-fat diet (Active Comparator): Participants will follow a high-fat diet. During the intervention phase, they will inoculate "Mutaflor Suspension" (E. coli Nissle 1917) (Single dose, 5 ml = 5x10^8 CFU).
  Blood samples, stool samples and clinical information will be collected during the study.
  Interventions: Drug: "Mutaflor Suspension" (E. coli Nissle 1917); Other: Blood samples; Other: Stool samples; Other: Clinical information
- Low-fat diet (Active Comparator): Participants will follow a low-fat diet. During the intervention phase, they will inoculate "Mutaflor Suspension" (E. coli Nissle 1917) (Single dose, 5 ml = 5x10^8 CFU).
  Blood samples, stool samples and clinical information will be collected during the study.
  Interventions: Drug: "Mutaflor Suspension" (E. coli Nissle 1917); Other: Blood samples; Other: Stool samples; Other: Clinical information

INTERVENTIONS:
Drug: "Mutaflor Suspension" (E. coli Nissle 1917) — Inoculation of "Mutaflor Suspension" (E. coli Nissle 1917)
  Other Names: Mutaflor Suspension
Other: Blood samples — Blood samples will be collected and analyzed at different study time points
Other: Stool samples — Stool samples will be collected and analyzed at different study time points
Other: Clinical information — Clinical information will be collected at different study time points using questionnaires

SUMMARY:
Recent experiments in the lab of Prof. WD Hardt revealed, that in mice, 24 h exposure to a high-fat diet results in a breakdown of colonization resistance against Salmonella typhimurium. Mechanistic experiments identified bile acids as the mediator for reduced colonization resistance. Exposure to a high fat diet leads to increased bile acid secretion which in turn modify the intestinal microbiota.

It is now the aim to verify the results of this study in human healthy volunteers. The nutritional habits of all participants will carefully be evaluated. In the intervention phase, participants will be exposed to either high-fat or low-fat diet and a controlled dose of the non-pathogenic bacteria E. coli Nissle. E. coli Nissle is the active compound for "Mutaflor®" and other probiotics.

It is planned to enumerate E. coli Nissle counts in the stool after Mutaflor ingestion and to quantify other changes of the human microbiota. The hypothesis is that a high-fat diet leads to increased bile acid secretion results in favorable growth conditions for E. coli Nissle, resulting in high bacterial counts in the stool.

DETAILED DESCRIPTION:
Infectious diarrhea causes substantial morbidity in Western countries and the developing world and leads to the use of considerable health resources. Antibiotic resistance continues to increase, potentially leading to a decrease in therapeutic options in the future. Important pathogens include Salmonella typhimurium (S. typhimurium) and pathogenic Escherichia coli (E. coli) which are genetically closely related.

The human intestine has considerable colonization resistance against bacterial pathogens. This resistance is largely mediated by the gut microbiota. Therefore, previous exposure to antibiotics or immunosuppression leading to a breakdown of the intestinal defense systems increase the risk for subsequent infection with S. typhimurium.

The composition of the human microbiome undergoes dramatic changes upon exposure to various factors including nutrition, physical activity, drugs and much more. Most studies focused on long-term exposure to various factors; however, since bacterial growth is rapid (doubling time of S. typhimurium under optimal conditions = 20min), even short-term variations in the environment could dramatically influence the human microbiota.

In the lab of Prof. WD Hardt, a mouse model of S. typhimurium enterocolitis has been established. Since most mouse strains are resistant against colonization with S. typhimurium, pretreatment with antibiotics is a requirement for induction of S. typhimurium enterolitis. However, recent experiments in the Hardt lab revealed, that in mice, 24 h exposure to a high-fat diet also results in a breakdown of colonization resistance, leading to Salmonella enterocolitis upon S. typhimurium infection. The same is true for E. coli strains. Subsequent experiments demonstrated that exposure to fatty acids is sufficient to overcome colonization resistance. Mechanistic experiments identified fat-elicited bile-release as the underlying mechanism: Exposure to a high fat diet leads to increased bile acid secretion; S. typhimurium can tolerate 10-fold higher bile acid concentrations than commensal bacterial, leading to a growth advantage of S. typhimurium compared to competing bacteria (WD Hardt et al., unpublished data).

The aim of this study is to verify the results of this study in human healthy volunteers. The nutritional habits of all participants will be carefully evaluated. In the intervention phase, participants will be exposed to either high-fat or low-fat diet and a controlled dose of the non-pathogenic bacteria E. coli Nissle. E. coli Nissle is the active compound for "Mutaflor®" and other probiotics. E. coli Nissle has therapeutic effects for the treatment of chronic inflammatory intestinal diseases. In contrast to other non-pathogenic E. coli strains, it exhibits a specific pattern of fitness factors but lacks prominent virulence factors. In vivo and in vitro experiments demonstrated both, protective effects against infection with intestinal pathogens as well as potent immunomodulatory properties. Growth of E. coli Nissle in the human gut resembles growth of S. typhimurium. Both bacteriae also share metabolic requirements for intestinal growth. Therefore, growth E. coli Nissle in the human intestine can be used as a marker for growth of E. coli strains, Salmonella typhimurium and related pathogens.

It is planned to enumerate E. coli Nissle counts in the stool after Mutaflor ingestion and to quantify other changes of the human microbiota. The hypothesize is that a high-fat diet, leading to increased bile acid secretion results in favorable growth conditions for E. coli Nissle, resulting in high bacterial counts in the stool.

The results of the study will help improving the understanding of the consequences of nutritional composition on the vulnerability of the human organism to bacterial infections. Such an improved understanding might enable designing preventive measures for the growth of unwanted E. coli strains (e.g. ESBL, pathogenic) or S. typhimurium infection and/ or a severe disease course and might ultimately help limiting antibiotic use and the evolution of antibiotic resistant pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Individuals free of abdominal complaints or symptoms
* Written informed consent
* Age 18 - 85 years
* Working at ETH Zurich or University of Zurich and trained and experienced in handling -80°C freezers at biosafety level 2.

Exclusion Criteria:

* Previous history of gastrointestinal disease or surgery (excludes appendectomy, hernia repair and surgery for anorectal disorders)
* Known diabetes mellitus, scleroderma, neurological impairment or other major diseases requiring ongoing management
* Immunesuppression
* Subjects with antibiotic therapy, proton pump inhibitors or laxatives within the last four weeks
* Pregnancy beyond week 12. "Mutaflor" intake is safe during pregnancy; however, special regulations are required to gain access to the -80°C freezers. No pregnancy test will be performed.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-24 (Estimated); Primary Completion 2019-09-24 (Estimated); Study Completion 2019-09-24 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration of E. coli Nissle bacteriae in all stool samples of each participant | 1, 2 and 5 days after E. coli Nissle inoculation
  Each participant's fecal samples will be analyzed for E. coli Nissle bacteriae. Only the stool samples acquired in intervention phase 1 will be considered. For each participant, the maximum concentration of E. coli Nissle in all stool samples (assessed by qPCR) will be used for the calculation of the primary outcome.
Comparison of E. coli Nissle concentration in feces between high-fat diet and low-fat diet | 1, 2 and 5 days after E. coli Nissle inoculation
  The concentration of E. coli Nissle bacteriae (CFU per g feces) in participants exposed to high-fat diet will be compared to the concentration of E. coli Nissle bacteriae in individuals exposed to low-fat diet (Mann-Whitney U test, a p-value <0.05 will be considered significant).

SECONDARY OUTCOMES:
Chemical composition of blood | Week 1 - 8
  For each participant's blood samples the chemical composition including bile acids, lipids, cholesterol and other compounds related to fat, cholesterol and bile acid metabolism will be determined (concentration, per μl blood). Samples at baseline, during intervention phase and the washout phase will be analyzed. For each compound the group exposed to low-fat diet and high-fat diet will be compared, respectively (intervention phase) or the group with the lowest and highest fat ingestion according to the nutritional protocol.
Chemical composition of stool | Week 1 - 8
  For each participant's stool samples the chemical composition including bile acids, lipids, cholesterol and other compounds related to fat, cholesterol and bile acid metabolism will be determined (concentration, per g stool). Samples at baseline, during intervention phase and the washout phase will be analyzed. For each compound the group exposed to low-fat diet and high-fat diet will be compared, respectively (intervention phase) or the group with the lowest and highest fat ingestion according to the nutritional protocol.
Microbiota composition: taxonomic composition | Week 1 - 8
  Same as 4, only the microbiota taxonomic composition in stool samples will be analyzed by ribosomal RNA gene sequencing. Analysis will also include tests for microbiota diversity (i.e. number of bacteria species identified). Findings will be compared to changes occurring in the microbiota of participants in the other study group.
Microbiota composition: metagenomic properties | Week 1 - 8
  Same as 4, only the metagenomic properties of the microbiota in stool samples will be analyzed by whole genome shotgun sequencing. Analyses will also test for metabolic pathways used by the microbiota. Microbiological and molecular biology methods will also be used to characterize bacteria strains associated with high-fat diet, low-fat diet and/ or changes in bile acid concentration.
Microbiota composition: E. coli content | Week 1 - 8
  Same as 4, only the E. coli content of stool samples will be analyzed by sequencing and conventional plating techniques. This will quantify E. coli Nissle and also all endogenous E. coli strains present in the sample.
Antibody response against E. coli Nissle | 3 weeks after inoculation of E. coli Nissle
  Antibody titers against E. coli Nissle will be determined by bacterial FACS or other appropriate techniques. Antibody titers at baseline, at 2 weeks and at 3 weeks will be determined. Individuals exposed to low-fat diet and high-fat diet will be compared. Measured variable: Antibody titers against E. coli Nissle and various E. coli strains.

CONTACTS AND LOCATIONS:
Overall Officials: Wolf-Dietrich Hardt, Prof. Dr., Principal Investigator — ETH Zurich, Institute of Microbiology
Locations (1):
- Institute of Microbiology (D-BIOL), ETH Zurich, Zurich, Switzerland